CLINICAL TRIAL: NCT04610554
Title: Lung Diffusing Capacity for Nitric Oxide and Carbon Monoxide Early After Mild-to-severe COVID-19
Status: Completed | Type: Observational
Sponsor: IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy (Other)
Responsible Party: Principal Investigator, Giovanni Barisione, MD - Chief, Respiratory Pathophysiology Unit, IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy
Other Study IDs: SARS-CoV-2_DLNO
Record Dates: First submitted 2020-10-29; First posted 2020-10-30 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: COVID-19 Pneumonia
Keywords: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Infection with severe acute respiratory syndrome-CoV-2 (SARS-CoV-2) may be associated with diffuse alveolar damage and pulmonary vasculitis. Thus, it is likely that pulmonary function changes may be seen in COVID-19 survivors. The aim of the present study was to test that simultaneously-determined lung diffusing capacity for nitric oxide and carbon monoxide may be useful to detect post-viral diffusive gas exchange abnormalities early after mild-to-severe COVID-19-related pneumonias.

DETAILED DESCRIPTION:
Infection with severe acute respiratory syndrome-CoV-2 (SARS-CoV-2) may be asymptomatic or associated with life-threatening interstitial pneumonia. Clinically, patients affected from severe coronavirus disease-19 (COVID-19) are described as exhibiting rapidly progressing acute respiratory failure with unusually low oxygen levels in arterial blood. On computed tomography scans, diffuse, peripheral "ground glass" opacities of the lung are seen while autopsy lung specimens showed diffuse alveolar damage and capillary endothelialitis.

The objective of the current study, conducted in patients who had recovered from mild-to-severe COVID-19 illness, was to test that simultaneously-determined lung diffusing capacity for nitric oxide (NO) and carbon monoxide (CO) may be of great use to early detect post-infective diffusive gas exchange abnormalities. More specifically, we hypothesized that measurement of membrane diffusive conductance for CO and pulmonary capillary volume may provide accurate information on residual changes of peripheral gas exchanging units of the lung related to previous SARS-CoV-2 infection.

ELIGIBILITY:
Inclusion Criteria:

* subjects were selected after two nasopharyngeal swabs negative for SARS-CoV-2

Exclusion Criteria:

* severe comorbidities potentially affecting pulmonary gas exchange

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: We collected the data of 74 Caucasian consecutive subjects admitted to hospital who had recovered from mild-to-severe COVID-19 and attended our laboratory as outpatients for follow-up purposes
Sampling Method: Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2020-05-14 (Actual); Primary Completion 2020-10-12 (Actual); Study Completion 2020-10-12 (Actual)

PRIMARY OUTCOMES:
Lung diffusing capacity for nitric oxide (DLNO) | At a time interval ranging from 15 to 189 days after two nasopharyngeal swabs negative for SARS-CoV-2
  Changes of DLNO after SARS-CoV-2 infection

SECONDARY OUTCOMES:
Lung diffusing capacity for carbon monoxide (DLco) | At a time interval ranging from 15 to 189 days after two nasopharyngeal swabs negative for SARS-CoV-2
  Changes of DLco after SARS-CoV-2 infection

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Barisione, MD, Principal Investigator — Sponsor should be IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy
Locations (1):
- IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Barisione G, Brusasco C, Garlaschi A, Baroffio M, Brusasco V. Lung diffusing capacity for nitric oxide as a marker of fibrotic changes in idiopathic interstitial pneumonias. J Appl Physiol (1985). 2016 May 1;120(9):1029-38. doi: 10.1152/japplphysiol.00964.2015. Epub 2016 Feb 18. PMID 26893034
- [Background] Barisione G, Bacigalupo A, Brusasco C, Scanarotti C, Penco S, Bassi AM, Lamparelli T, Garlaschi A, Pellegrino R, Brusasco V. Mechanisms for reduced pulmonary diffusing capacity in haematopoietic stem-cell transplantation recipients. Respir Physiol Neurobiol. 2014 Apr 1;194:54-61. doi: 10.1016/j.resp.2014.01.018. Epub 2014 Feb 1. PMID 24495442
- [Result] Barisione G, Garlaschi A, Occhipinti M, Baroffio M, Pistolesi M, Brusasco V. Value of lung diffusing capacity for nitric oxide in systemic sclerosis. Physiol Rep. 2019 Aug;7(13):e14149. doi: 10.14814/phy2.14149. PMID 31264386
- [Derived] Barisione G, Brusasco V. Lung diffusing capacity for nitric oxide and carbon monoxide following mild-to-severe COVID-19. Physiol Rep. 2021 Feb;9(4):e14748. doi: 10.14814/phy2.14748. PMID 33625799